CLINICAL TRIAL: NCT03142867
Title: The Prevalence of Nonalcoholic Fatty Liver Disease (NAFLD) in Adults
Acronym: PREV
Status: Terminated | Type: Observational
Why Stopped: Study complete but no analysis, publications or presentations of any collected data will be performed. Investigator left the site and study was halted.
Sponsor: The Geneva Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20513
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis
Keywords: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis; Prevalence; Coronary Artery Disease; PDFF
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An additional 5 ml of whole blood and 5 ml of serum will be collected and stored by a research coordinator, nurse, research assistant, or investigator for analysis of specific biomarkers to include Hyaluronic acid, CK-18 (M30), FGF-21, Mac-2BP, FAS, AFP, YKL-40, Alpha-2-macroglobulin and a panel of 46 fatty acids during the liver biopsy appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: The target population for this study is male and female patients (age 18 to 80) and will consist of retired and active military personnel and their dependents. There will be no race, ethnic, or gender limitations to enrollment.
  The control group will be made of individuals who do not meet the qualifications for a liver biopsy.
  Interventions: Other: non-applicable
- NAFLD: The target population for this study is male and female patients (age 18 to 80) and will consist of retired and active military personnel and their dependents. There will be no race, ethnic, or gender limitations to enrollment.
  The NAFLD group will be made of individuals who qualify for a liver biopsy and have histologically proven NAFLD.
  Interventions: Other: non-applicable
- NASH: The target population for this study is male and female patients (age 18 to 80) and will consist of retired and active military personnel and their dependents. There will be no race, ethnic, or gender limitations to enrollment.
  The NASH group will be made of individuals who qualify for a liver biopsy and have histologically proven NASH.
  Interventions: Other: non-applicable

INTERVENTIONS:
Other: non-applicable — non-applicable

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a global health concern with a suspected increasing prevalence due to the rise in obesity and diabetes mellitus. The vast majority of patients will have isolated steatosis or steatosis with mild inflammation that is very unlikely to progress in severity. However, about 25% of patients with NAFLD have non-alcoholic steatohepatitis (NASH), the more aggressive form of the disease that is associated with fibrosis progression and potential risk for cirrhosis and end-stage liver disease complications. Additionally, multiple studies have demonstrated an association between NAFLD and the presence of coronary artery disease by either coronary CT angiography (CCTA) or coronary artery calcium (CAC) score. Cardiovascular disease is the most important cause of mortality in patients with the entire spectrum of NAFLD. In the era of advanced imaging and functional vascular assessment it is possible that novel risk assessments are poised to refine overall prognostic estimation in this population. Multiple analyses have suggested that NAFLD is an independent and strong predictor of significant CAD independent of cardiovascular risk factors, including a significant burden of high risk CCTA findings in one analysis of symptomatic patients in the emergency department. Given the multiple metabolic derangements inherent in the NAFLD population, endothelial dysfunction is also an important contributor to global cardiovascular dysfunction. Furthermore, data suggests that patients with NAFLD may be at increased risk of adenomatous polyp formation and colorectal adenocarcinoma. In addition, it is suboptimal to require a liver biopsy to diagnose NASH. Recent imaging advances have made it possible to assess liver fibrosis but have yet to be fully studied in NAFLD. The purpose of this study is to assess the current prevalence and severity of NAFLD in adult subjects. Secondary endpoints include correlation to new vascular function (cine scan of the abdominal aorta) and echocardiographic imaging modalities available at BAMC and to circulating biomarker panels as well as to determine the prevalence and severity of CAD by multidetector coronary CT angiography with subject outcomes being monitored prospectively. Additionally, correlation of NAFLD diagnosis to colonoscopy findings will be performed.

DETAILED DESCRIPTION:
In this prospective study, adult patients ranging in age from 18-80, routinely seen in the Brooke Army Medical Center Gastroenterology clinics will be eligible for enrollment. Approximately 950 adult patients will be enrolled. In phase I the prevalence of NAFLD and NASH will be determined, non-invasive imaging techniques for the diagnosis of NAFLD and NASH will be explored, and the relationship between colon polyps and NAFLD will be evaluated. Phase II will be offered to participants that qualified for a liver biopsy. In phase II the prevalence and severity of CAD, endothelial dysfunction, and diastolic dysfunction within the population of subjects with NAFLD will be determined.

Phase I:

After obtaining informed consent and confirming that the subject has met inclusion and exclusion criteria for the study, the study will employ a questionnaire to be completed by the subject. This questionnaire will include data such as race and ethnic group, past medical history, current medications, etc. The subject will then have routine labs (liver function tests, fasting insulin, glucose, and a pregnancy test for all female subjects), FibroScan® and MRE/MRI done to assess for the presence or absence of hepatic steatosis, inflammation, fibrosis, iron quantification and diameter and luminal characteristics of the abdominal aorta. Subjects will be called by the PI or an AI to return to the clinic for additional study procedures to include a core liver biopsy if they are identified to have one or more of the following:

* greater or equal to 5% steatosis on MRI or
* liver stiffness greater than 7 kPa on Fibroscan®, or
* evidence of fibrosis on MRE or
* LIF score of 2.0 or greater

The PI/AI will let the subject know that he/she qualifies for further diagnostic testing as part of the trial and will discuss tests results with them in detail.

FibroScan examination will be performed to assess liver stiffness according to the manufacturer's recommendation and in accordance with the device's FDA clearance. The device is equipped with two probes (M and XL) dedicated to different morphology and operating at different measurement depths. The M probe operates between 25 and 65 mm below the skin surface and the XL probe operates between 35 and 75 mm. The device's software automatically recommends which probe is the most appropriate during examination based on the real time assessment of the skin to liver capsule distance (automatic probe selection tool). The FibroScan used in this study will be equipped with a software allowing, in addition to liver stiffness, measurement of the Controlled Attenuation Parameter (CAP) which is related to liver steatosis with different algorithm. This additional software feature is FDA approved. Operators will be trained and certified by the manufacturer or its local representative. Recommendation from the Automatic Probe Selection tool will be followed. At least ten valid measurements should be obtained. De-identified acquisition files will be reviewed by the device's manufacturer (Echosens) to confirm the operator's choice of measurement depths and eventually change them as well as analyze the additional ultrasonic signals.

In addition to the Fibroscan, a second non-invasive imaging technique, MRE/MRI Liver MultiScan for detecting steatosis, inflammation and liver fibrosis or stiffness will be conducted. This data will be used to correlate with the presence of NAFLD/NASH. MRI-Liver MultiScan is a post MRI processing software. It involves a specialized magnetic resonance imaging (MRI) technique/sequences that measures fat, iron and fibrosis in the liver using T1 mapping. The procedure has no need for intravenous contrast. LiverMultiScan is currently approved by the FDA for use with Siemens 3T MRI with E11 software. However, this MRI model is not being used at BAMC. Therefore, the use of LMS locally will conducted under an IDE exemption for diagnostic devices (21 CFR 812.2(c))(3). The LMS software will not be used to clinically diagnose subjects. Rather, data will be collected and analyzed by the site and manufacturer (Perspectum) with the knowledge that MRI is not performed in accordance with LMS labeling.

BAMC Radiology will work in collaboration with Perspectum to complete the post processing review of the MRI image data to correlate with the presence of NAFLD/NASH. The BAMC Radiology Department AI's will de-identify the image data (remove all PHI), load on a secure server and have Perspectum Diagnostics complete the post-processing interpretations.

The MR elastography scan will be conducted in conjuncture with the MRI scan and post-processed by AIs within the BAMC Radiology Department. In addition, AIs in the BAMC Radiology Department will conduct a safety read of all scans. The results of the MRE and the safety read will be placed in the subject's electronic medical record.

Participants that qualify for a core liver biopsy based upon the results from the FibroScan and MRE/MRI LiverMultiScan will be asked to return to specimen collection for additional blood work prior to the liver biopsy. This will consist of a complete blood count (CBC), coagulation panel, fasting lipid panel, GGT, vitamin D level, renal function panel, ferritin, hemoglobin A1C, and chronic hepatitis panel.

Subjects will then undergo a percutaneous liver biopsy to establish diagnosis of NASH. This will occur in the Gastroenterology Clinic at Brooke Army Medical Center. The liver tissue will be submitted to BAMC Pathology Department for evaluation by an AI, an experienced hepatopathologist. The pathology results will be used to identify subjects who have the more severe form of NAFLD, NASH. The pathologist will provide an overall diagnostic interpretation based on the criteria reported by Brunt et al. and by the NAFLD Activity Score (NAS). According to this scoring system, the degree of steatosis and inflammatory activity is measured using a zero to eight scale (steatosis=0-3; lobular inflammation=0-3; ballooning=0-2). The NAS is the unweighted sum of steatosis, lobular inflammation, and hepatocellular ballooning scores. The stage of fibrosis will be assessed using a zero to four scale (0=no fibrosis; 1=mild/moderate zone three perisinusoidal fibrosis, or portal/periportal fibrosis only; 2= perisinusoidal and portal/periportal fibrosis; 3= bridging fibrosis; 4= cirrhosis). Additionally, at the time of liver biopsy, 4 additional unstained slides will be prepared for morphometry analysis by Echosens. The liver histological diagnosis will be established by an experienced pathologist blinded to the clinical characteristics of the subjects, radiographic studies and the serum biomarkers. The outside expert pathologist will use the same scoring system as the local pathologist. If there is a discrepancy between the two pathology results for a subject the final determination will be made by the local BAMC pathologist. An addendum will be placed in the electronic medical record by the BAMC pathologist. The subject will be informed of the change and documentation of the new diagnosis and any further treatments will be made in AHLTA.

Echosens will use the liver biopsy slides to correlate the FibroMeter™ NAFLD/VCTE test with liver fibrosis and the presence of NAFLD and NASH. FibroMeter™ is a non-invasive diagnostic test that evaluates the level of fibrosis in the liver using patient clinical data (age and weight) and a proprietary selection of standard clinical lab results including platelets, AST, ALT, ferritin, glucose and Alpha-2-macroglobulin levels. The results of these locally run tests will be entered into the Echosens FibroMeter website for FibroMeter NAFLD/VCTE calculation. This test is approved in Europe and provides means for detection of significant fibrosis, detection of cirrhosis (screening for esophageal varices and hepatocellular carcinoma) and a quantitative estimate of fibrosis staging, thereby providing opportunity for serial monitoring of fibrosis in suspected cases. The FibroMeter test result will then be used by Echosens to correlate with the morphometry analysis. All results are identified with only the subject study number. Results from the FibroMeter test will not be used to support a FDA marketing application. Additionally, the results of the FibroMeter will not be used clinically nor to determine the performance of any subsequent research procedure. The results will not be placed in the subject's medical records.

An additional 5 ml of whole blood and 5 ml of serum will be collected and stored by a research coordinator, nurse, research assistant, or investigator for analysis of specific biomarkers to include Hyaluronic acid, CK-18 (M30), FGF-21, Mac-2BP, FAS, AFP, YKL-40, Alpha-2-macroglobulin and a panel of 46 fatty acids during the liver biopsy appointment. Phlebotomies will be performed in Hepatology Research. The stored serum will be kept in the BAMC Gastroenterology Clinic in a -80 degree freezer and batch shipped to an outside lab periodically for analysis. Specimens will be identified by a designated research code only available to the local study team, thereby removing any personal identifiers on specimens prior to shipment to an outside lab.

In order to address aim 3, subjects enrolled in the study who have undergone or will undergo colonoscopy during study participation as part of their routine clinical care will have their AHLTA/CHCS records reviewed and those with colon polyps or colon masses will be evaluated against their imaging study findings. The correlation between colon polyp number/severity and the presence of NAFLD will be ascertained.

Subjects qualifying for a liver biopsy will be referred to the study team members in the Cardiology clinic with the option to enroll in Phase II of the protocol.

Phase II:

Phase II will consist of three cardiology procedures.

1. Coronary CT angiography: All subjects who meet inclusion criteria for a percutaneous liver biopsy, are consented to phase II, and do not have known CAD defined as prior percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) or have not undergone CCTA within the previous 12 months, will undergo a CCTA with CAC score. Subjects undergoing this portion of the analysis will need a renal function panel within 30 days of the scan date with a glomerular filtration rate (GFR) of ≥ 60 mls/min/1.73m2 by the Cockcroft-Gault equation, no prior history of an allergic reaction to intravenous CT contrast, and no contraindications to administration of sublingual nitroglycerin and nodal blocking agents. All CCTA scans will be analyzed by a cardiologist with level III ACC/ACR certified imaging expertise in accordance with the Society of Cardiovascular Computed Tomography (SCCT) guidelines. Scans will be performed in accordance with SCCT guidelines. Studies will be obtained utilizing a 128-slice dual source scanner with a high pitch, single heart beat image acquisition capabilities (Somatom Definition Flash CT®, Siemens, Erlagen, Germany). CAC scanning will occur first at a standard tube voltage of 120 keV and 3 mm slice acquisition and CareDose® modulation of tube current enabled for all scans. CT technologist will be responsible for contacting the on-call CT imaging specialist for CAC score ≥400 prior to proceeding to CCTA acquisition. Continuation to CCTA will be at the discretion of the CT imaging specialist. Tube voltage and image acquisition protocoling will be selected by the CT technologist in consultation with the on-call cardiac CT imaging specialist in accordance with the flowsheet depicted in Appendix 3. Tube voltage of 120keV will be used for BMI > 30 and lowered to 100keV for BMI ≤ 30. CareDose® modulation of tube current will be enabled for all scans. Pretreatment with nodal blocking agents will be as follows: for HR < 70 bpm and systolic blood pressure (SBP) > 100 mm Hg will be given 50mg orally, for HR > 70 bpm and SBP > 100 mm Hg will be given 100mg orally, and nodal blocker will be held for patients with HR < 50 bpm or SBP < 100 mm Hg at the time of evaluation. Additional nodal blocker will be administered following initial dosing at the discretion of the cardiac imaging specialist. All subjects with SBP > 90 mm Hg and without a history of phosphodiesterase inhibitor usage in the preceding 72 hours received nitroglycerin spray 0.4-0.8 mg within 2 minutes of scan acquisition. High-pitched, prospective, ECG-triggered helical scanning will be performed with heart rate (HR) < 60 bpm and HR variability < 5 beats or with HR < 60 bpm at the discretion of the imaging specialist. The remaining scans will be performed using prospective, ECG triggering acquisition centered at 70%-phase with between 10-20% padding (40-80% of the R-R interval). Visapaque® intravenous (IV) contrast will be used for all scans. A triphasic injection protocol consisting of 75mL of IV contrast followed by 40 mL of 50% contrast mixed with normal saline chased with normal saline at a flow rate of 5 mL/second will be used for all scans with total IV contrast volume of 105-125 mL. Contrast flow rates will be increased to 6 ml/second for patients with BMI > 30. Coronary artery stenosis by CCTA will be determined on a per-patient and per-vessel basis using an 18 segment model in accordance with SCCT guidelines for interpretation. The major epicardial coronary arteries (left main, left anterior descending, left circumflex, and right coronary arteries) will be graded for severity of CAD, defined as obstructive CAD (>50% stenosis), non-obstructive CAD (≤50% stenosis), or no CAD (vessels free of angiographic evidence of disease), respectively. The posterior descending artery will be included in the left circumflex or right coronary artery groups depending on its origin. The subject will have the option of declining the CCTA and CAC scan. Subjects with known CAD as defined on recent prior CCTA (within last 12 months) will not undergo CCTA, but their CAD history and/or prior CCTA results will be included in the analysis.
2. Transthoracic Echocardiography (TTE): All subjects who meet inclusion criteria for a percutaneous liver biopsy and consented to phase II will undergo an assessment of cardiovascular diastolic performance measured using 2D and 3D transthoracic echocardiography (TTE) with Doppler technology. The TTE will be performed during a scheduled outpatient time slot at the convenience of the patient.
3. EndoPAT: Endothelial function will be measured in subjects who qualify for liver biopsy and consent to phase II using the EndoPAT 2000®.. Every effort will be made to conduct the EndoPat test on the same day as the CCTA for subject convenience. The EndoPAT 2000® uses digital pulse amplitude tonometry. The EndoPAT device comprises a pneumatic plethysmograph that applies uniform pressure the surface of the distal finger. Throughout the test, the inflation pressure of the device will be set at 10 mmHg below the diastolic blood pressure or 70 mmHg, whichever is lower. Baseline pulse amplitude measurements will be taken for 5 minutes. Arterial flow will then be transiently interrupted by inflating a pneumatic cuff placed on the patient's forearm. The cuff will be inflated to 200 mmHg or 60 mmHg plus the systolic blood pressure, whichever is higher. The pulse amplitude will be recorded for 5 minutes during the occlusion phase. The blood pressure cuff is then deflated and post test measurements are recorded for 5 additional minutes. Pre and post test pulse amplitudes are compared to assess the degree of reactive hyperemia.

Subjects found to have evidence of coronary artery calcium, endothelial dysfunction, diastolic dysfunction and/or presence of non-calcific atherosclerosis on CCTA with maximal stenosis < 50% will be referred to the cardiology clinic for assessment of cardiovascular risk and aggressive medical and lifestyle risk factor modification. Patients with stenosis ≥ 50% will also be referred to the cardiology clinic to be evaluated further for the need for additional ischemic testing at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Phase I:

  1. Male and female patients (≥18 years of age to 80)
  2. Eligible for care at Brooke Army Medical Center

Phase II:

1. Met the criteria for qualification for a percutaneous liver biopsy and completed Phase I
2. Eligible for care at Brooke Army Medical Center

Exclusion Criteria:

* Phase I:

  1. Patients with excessive alcohol use will be excluded as defined as >21 units of alcohol/week for men and 14 units of alcohol/week for women over a 2 year time frame. One drink "unit" or one standard drink is equivalent to a 12-ounce beer, a 4-ounce glass of wine, or a 1-ounce shot of hard liquor.
  2. Patients with prior history of liver disease to include chronic hepatitis B or C, hemochromatosis, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, HIV, or prior documentation of NAFLD.
  3. Patients on medications known to cause fatty liver disease: tamoxifen, corticosteroids, amiodarone, methotrexate, valproic acid
  4. Patients carrying an implantable active medical device such as a pacemaker or a defibrillator
  5. Pregnant women

Phase II:

1. CCTA/CAC only: GFR <60 mls/min/1.73m2 or IV contrast dye allergy
2. CCTA/CAC only: contraindications to atrioventricular (AV) nodal blocking agents (high degree AV block without permanent pacemaker, asthma, allergy to nodal blocking agents).
3. Known CAD defined as previous PCI or CABG (Note: Subjects with CCTA within the past 12 months will not be excluded from study and repeat scan will not be needed but the results of that previous scan will be included in the prevalence and severity analysis.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will include all adults presenting to the BAMC Gastroenterology clinic.
  The target population for this study is male and female patients (age 18 to 80) and will consist of retired and active military personnel and their dependents. BAMC is the only study site. There will be no race, ethnic, or gender limitations to enrollment.
Sampling Method: Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of NAFLD | from the date of consent to the completion of phase I (up to 3 months)
  Determine the prevalence of NAFLD in military beneficiaries between ages 18 to 80. This will be determined by the % of subjects determined to have NAFLD via liver biopsy.
Prevalence of NASH | from the date of consent to the completion of phase I (up to 3 months)
  Determine the prevalence of NASH in military beneficiaries between ages 18 to 80. This will be determined by the % of subjects determined to have NASH via liver biopsy.

SECONDARY OUTCOMES:
proton density fat fraction | Determined at the date of MRI (1 day)
  % fat in the liver determined via MRI and LiverMultiScan software
Liver stiffness measure by Fibroscan | Determined at the date of Fibroscan (1 day)
  Liver stiffness will be determined via kPa value from Fibroscan
Liver stiffness measure by MRE | Determined at the date of MRE (1 day)
  Liver stiffness will be determined via kPa value from MRE
Stages of fibrosis and grades of steatosis | determined at the date of liver biopsy tissue evaluation (1 day)
  determined by a pathologist reading liver biopsy slides and Brunt scoring system
Prevalence of colon polyps | determined at the date of colonoscopy (1 day)
  Determine the prevalence and severity of colon polyps within the population of subjects identified as having NAFLD and correlate these findings to those without NAFLD.
Prevalence and severity of CAD | determined at the date of CCTA (1 day)
  Determine the prevalence and severity of CAD by CCTA and CAC scoring within the population of subjects identified as having NAFLD. Prospectively follow patients undergoing CCTA/CAC scoring for major cardiovascular events (myocardial infarction, stroke/TIA, coronary revascularization, or death).
Prevalence and severity of endothelial dysfunction with peripheral tonometry | determined at the date of the EndoPat Test (1 day)
  Determine the prevalence and severity of endothelial dysfunction with peripheral tonometry within the population of subjects identified as having NAFLD. Prospectively follow patients undergoing with peripheral tonometry for major cardiovascular events (myocardial infarction, stroke/TIA, coronary revascularization, or death).
Prevalence of diastolic dysfunction | determined at the date of the transthoracic echocardiogram (1 day)
  Determine the prevalence of diastolic dysfunction with transthoracic echocardiography within the population of subjects identified as having NAFLD

CONTACTS AND LOCATIONS:
Overall Officials: Angelo H Paredes, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- San Antonio Military Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dennis A, Kelly MD, Fernandes C, Mouchti S, Fallowfield JA, Hirschfield G, Pavlides M, Harrison S, Chakravarthy MV, Banerjee R, Sanyal A. Correlations Between MRI Biomarkers PDFF and cT1 With Histopathological Features of Non-Alcoholic Steatohepatitis. Front Endocrinol (Lausanne). 2021 Jan 27;11:575843. doi: 10.3389/fendo.2020.575843. eCollection 2020. PMID 33584535